CLINICAL TRIAL: NCT06738836
Title: An Open-Label Phase 1 Study in Healthy Male Subjects to Investigate the Absorption, Metabolism and Excretion of [14C]-EDG-7500 Following Single-Dose Oral Administration
Brief Title: A Study to Evaluate the Absorption, Metabolism, And Excretion Of Orally Administered [14C]-EDG-7500
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Edgewise Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EDG-7500-104
Record Dates: First submitted 2024-12-04; First posted 2024-12-18 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Human AME (Experimental)
  Interventions: Drug: [14C]-EDG-7500

INTERVENTIONS:
Drug: [14C]-EDG-7500 — Oral liquid suspension

SUMMARY:
The purpose of this study is to:

1. Assess the mass balance (i.e., the cumulative elimination of 14C-related material in urine and feces, compared to the administered amount of radioactive isotope) of [14C]-EDG-7500 following a single oral dose of EDG-7500 containing a radioactive tracer, in healthy, adult male subjects.
2. Characterize the pharmacokinetics of EDG-7500 in plasma and of 14C-related material in whole blood, plasma, urine and feces following a single oral dose of EDG-7500 containing a radioactive tracer, in healthy, adult male subjects.

ELIGIBILITY:
Key Inclusion Criteria:

* Biological males ≥ 18.0 and < 55.0 years of age at time of providing Informed Consent.
* Body mass index (BMI) ≥ 18.0 kg/m2 and ≤ 32.0 kg/m2 at Screening; body weight ≥ 55.0 kg and ≤ 100.0 kg at Screening.
* Subjects with female sexual partner(s) of reproductive potential may be enrolled if the male:

  1. is documented to be surgically sterile (i.e., successfully vasectomized); or
  2. agrees to use double-barrier contraception for at least 3 months after receiving study drug and agrees to refrain from sperm donation from the time of Screening through 3 months post dose.
* Negative for hepatitis B surface antigen, hepatitis C virus antibody and human immunodeficiency virus antibody and antigen.
* Non-smoker

Key Exclusion Criteria:

* Clinically significant abnormal medical history, or any abnormal findings on physical examination, vital signs, ECG or laboratory tests at Screening, Admission or predose on Day 1.
* Any history of serious allergic/hypersensitivity reactions.
* History or presence of alcohol or drug abuse within 2 years prior to Screening.
* Recent history of incomplete bladder emptying with voiding or awakening more than once at night to void. Usual habit of < 1 or > 3 bowel movements per day.
* Exposure to radiation for therapeutic or diagnostic reasons (except dental X rays and plain X rays of the thorax and bony skeleton) within the past 12 months .
* Participation in another clinical study in which a [14C]-labeled drug was administered within 1 year prior to Admission.
* QTcF interval (QT interval corrected for heart rate per Fridericia's formula) > 450 msec at Screening, Admission or predose on Day 1. Personal and family history of long QT syndrome or unexplained sudden death in a first-degree relative under 50 years of age.
* Glomerular filtration rate (GFR) < 80 mL/min/1.73 m2
* Loss or donation of blood (approximately 500 mL or greater) within 60 days prior to study drug administration on Day 1; donation of bone marrow or peripheral stem cells within 90 days prior to study drug administration on Day 1; or donation of plasma within 30 days prior to study drug administration on Day 1.

Additional protocol defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2024-12-03 (Actual); Primary Completion 2025-01-17 (Actual); Study Completion 2025-01-17 (Actual)

PRIMARY OUTCOMES:
Mass Balance | From Day -1 through study completion (up to 19 days)
Pharmacokinetics of EDG-7500 in plasma and 14C total radioactivity in plasma and whole blood as measured by Cmax | From Day 1 to study completion (up to 18 days)
Pharmacokinetics of EDG-7500 in plasma and 14C total radioactivity in plasma and whole blood as measured by Tmax | From Day 1 to study completion (up to 18 days)
Pharmacokinetics of EDG-7500 in plasma and 14C total radioactivity in plasma and whole blood as measured by T1/2 | From Day 1 to study completion (up to 18 days)
Pharmacokinetics of EDG-7500 in plasma and 14C total radioactivity in plasma and whole blood as measured by AUC0-inf | From Day 1 to study completion (up to 18 days)

SECONDARY OUTCOMES:
Metabolite profile | From Day -1 through study completion (up to 19 days)
Safety as measured by occurrence of adverse events, clinical laboratory evaluations, 12-lead ECG and vital sign measurements | From screening through study completion (up to 54 days)

CONTACTS AND LOCATIONS:
Locations (1):
- Pharmaron Clinical Pharmacology Center, Inc., Baltimore, Maryland, United States